CLINICAL TRIAL: NCT02321462
Title: Efficacy, Safety and Tolerability of a Split-dose of a New Bowel Cleansing Preparation (Eziclen) in Adult Subjects Undergoing Colonoscopy: A Phase III, Multicentre, Randomised, 2 Parallel Group, Comparative Versus Fortrans®, Non-inferiority, Investigator-blinded Study
Brief Title: Efficacy, Safety and Tolerability of Eziclen in Adult Subjects Undergoing Colonoscopy
Acronym: ESTOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: A-38-58800-002
Record Dates: First submitted 2014-12-17; First posted 2014-12-22 (Estimated); Results first posted 2019-02-27 (Actual); Last update posted 2019-03-04 (Actual); Status verified 2019-03

CONDITIONS: Bowel Cleansing
Keywords: preparation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Eziclen (Experimental)
  Interventions: Drug: Eziclen
- Fortrans® (Active Comparator)
  Interventions: Drug: Fortrans®

INTERVENTIONS:
Drug: Eziclen — Eziclen solution administered orally as split-dose the day before and on the day of colonoscopy.
  Arms: Eziclen
Drug: Fortrans® — Fortrans® solution administered orally as split-dose the day before and on the day of colonoscopy.
  Arms: Fortrans®

SUMMARY:
The purpose of this study is to demonstrate that Eziclen is non-inferior to Fortrans® (the reference colonic lavage in Russia) administered in adult subjects scheduled to undergo colonoscopy for a routinely accepted diagnostic indication.

ELIGIBILITY:
Inclusion Criteria:

* Provision of written informed consent signed prior to any study related procedures
* Male or female, at least 18 years old undergoing colonoscopy for a routine diagnostic indication:

  1. Routine cancer screening
  2. Polyp or neoplasm history
  3. Diagnostic procedure for occult bleeding or anaemia
  4. Diarrhoea or constipation of unknown aetiology
  5. IBD if not in severe acute phase
  6. Abnormal ultrasound exam (i.e. mass in abdomen)
  7. Evaluation of barium enema or computed tomography (CT) scan results
* In good clinical condition (physical exam and medical history)
* Subjects with an adequate fluid balance, and adequate electrolyte balance (measured during screening K, Na, Cl, bicarbonate within normal/near normal range)

Exclusion Criteria:

* Has abnormal baseline findings, any other medical condition(s) or laboratory findings that, in the opinion of the investigator, might jeopardise the subject's safety or decrease the chance of obtaining satisfactory data needed to achieve the objective(s) of the study.
* Has an advanced carcinoma or any other colon disease leading to excessive mucosal fragility.
* Has a known or suspected gastrointestinal (GI) obstruction, gastric retention, gastroparesis, or disorder of gastric emptying.
* Has a known or suspected ileus.
* Has a bowel perforation.
* Has profuse vomiting.
* Needs a therapeutic procedure (e.g. polypectomy, mucosectomy).
* Has toxic colitis or megacolon.
* Is in severe acute phases of active IBD, as a contraindication for colonoscopy.
* Has acute GI bleeding.
* Underwent previous GI surgeries (e.g. colostomy, colectomy, gastric bypass, stomach stapling).
* Has impaired consciousness predisposing to pulmonary aspiration.
* Needs a colonoscopy for foreign body removal and decompression.
* Underwent previous incomplete colonoscopy.
* Has a known severe renal insufficiency (glomerular filtration rate (GFR) <30 mL/min/1.73 m2).
* Has a known severe liver insufficiency (Child-Pugh grade C: 10 to 15 points).
* Suffers from uncorrected dehydration.
* Has ascites.
* Suffers from severe congestive heart failure (classes III and IV).
* Has hyperuricemia with clinical manifestation as gouty arthritis.
* Is pregnant or lactating.
* Is a female at risk of pregnancy and not using an acceptable contraceptive method during the study. Females of childbearing potential must provide a negative pregnancy test at start of study and must be using oral, double barrier (condom with spermicidal jelly, foam suppository, or film; diaphragm with spermicide; or male condom and diaphragm with spermicide), or injectable contraception or an intra-uterine device. Nonchildbearing potential is defined as postmenopause for at least one year, surgical sterilisation or hysterectomy at least three months before the start of the study.
* Has any known hypersensitivity to the active substances or to any of the preparation excipients (Eziclen or Fortrans®: polyethylene glycol (PEG) (macrogol), sodium sulphate, potassium sulphate, magnesium sulphate, sodium chloride, potassium chloride, sodium bicarbonate, sucralose, sodium saccharin, sodium benzoate, citric acid, malic acid, and fruit cocktail flavor).
* Patient has any mental condition rendering the subject unable to understand the nature, scope and possible consequences of the study, and/or evidence of an uncooperative attitude
* Patient was treated with any other IMP within the last 30 days before study entry
* Patient is likely to require treatment during the study with drugs that are not permitted by the study protocol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 296 (Actual)
Dates: Start 2015-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (3):
- Russia (3):
  - State Healthcare Institution Municipal Clinical Hospital No. 31 of Moscow, Moscow
  - Federal State Budgetary Institution "State Scientifical Center of Coloproctology", Moscow
  - State Healthcare Institution of Yaroslavl Region "Regional Clinical Cancer Hospital", Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Adult patients due to undergo colonoscopy for a routine diagnostic indication were enrolled into this noninferiority phase 3 study at 3 study centres in Russia. First patient started: 13 March 2015; last patient completed: 28 December 2015.
Pre-assignment Details: 305 patients were screened for inclusion, and 296 patients met all inclusion criteria and none of the exclusion criteria and were randomised to treatment. 294 patients received study treatment, and 2 patients were excluded from the safety and intention-to-treat (ITT) populations as they did not receive study treatment prior to colonoscopy.
Groups:
- Eziclen: Patients were randomised to receive an oral split-dose of Eziclen on Day 1 and Day 2. The first dose was taken the evening of Day 1 before the colonoscopy and the second dose was taken 10 - 12 hours after the evening dose on the day of the colonoscopy. Colonoscopy was performed on Day 2, at least 1 hour and no more than 6 hours after the last dose of Eziclen.
- Fortrans®: Patients were randomised to receive an oral split-dose of Fortrans® on Day 1 and Day 2. The first dose was taken the evening of Day 1 before the colonoscopy and the second dose was taken 10 - 12 hours after the evening dose on the day of the colonoscopy. Colonoscopy was performed on Day 2, at least 3 hours and no more than 6 hours after the last dose of Fortrans®.
Period: Overall Study
Arm/Group | Eziclen | Fortrans®
Started (Patients randomized to each arm) | 147 | 149
ITT Population (Patients assessed according to their randomised treatment, regardless of treatment they received) | 146 | 148
Treated Patients (Patients assessed according to actual treatment they received (See Limitations and Caveats section)) | 147 | 147
Safety Population (Patients assessed according to actual treatment they received (See Limitations and Caveats section)) | 147 | 147
Completed | 141 | 146
Not Completed | 6 | 3
Not completed — Withdrawal by Subject | 5 | 2
Not completed — Subject withdrawn before any treatment | 1 | 1

BASELINE CHARACTERISTICS:
Population: The safety population consisted of all randomised patients who received even a partial dose of study treatment. Patients were analysed according to the actual treatment received.
Arm/Group | Eziclen | Fortrans® | Total Title
Number analyzed (Participants) | 147 | 147 | 294
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.6 (13.0) | 54.0 (13.0) | 53.8 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 108 | 105 | 213
  Male | 39 | 42 | 81

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Percentage of Patients With Successful Overall Colon Preparation, Assessed by the Global Score of the Boston Bowel Preparation Scale (BBPS).
Description: The BBPS score for each colon segment (right, transverse and left colon) was assessed by 3 blinded experts as follows: 0=unprepared segment with mucosa not seen due to solid stool that cannot be cleared , 1=portion of mucosa of the segment seen, but other areas not well seen due to staining, residual stool and/or opaque liquid, 2=-minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of segment seen well, 3=entire mucosa of segment seen well with no residual staining, small fragments of stool and/or opaque liquid.
  A reconciled score based on the 3 blinded reviews was used to calculate the global BBPS score, ranging from 0 to 9 (worst to best). A successful overall colon preparation was defined as a global score ≥6 for the 3 colon segments.
  The percentage of patients with a successful preparation was determined using a logistic regression model, adjusted on centre, age class (<= 65; > 65), gender and inflammatory bowel disease (IBD) status.
Time Frame: Colonoscopy was performed on Day 2.
Population: The per protocol (PP) population consisted of all randomised patients who received the preparation of study treatment (complete or partial), who underwent the colonoscopy procedure and for whom no major protocol violation occurred until colonoscopy. Patients were assessed according to the randomised treatment, regardless of treatment received.
Measure: Number (95% Confidence Interval); unit: Adjusted percentage of patients
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 139 | 135
Adjusted percentage of patients | 97.18 [89.48 to 99.29] | 97.65 [90.67 to 99.44]
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; A multivariate logistic regression model, adjusted on centre, age class (≤65; >65), gender and IBD status (No IBD, IBD) was used; Test type: Non-Inferiority — Non-inferiority would be demonstrated if the lower limit of the 95% confidence intervals (CI) of the difference was higher than the predefined noninferiority margin (-15%); Adjusted difference = -0.46, 95% CI 2-sided [-4.22 to 3.29] — To investigate noninferiority of Eziclen compared to Fortrans®, the adjusted difference between these 2 groups was calculated with 95% CI of the adjusted difference

2. Secondary Outcome: Mean BBPS Score by Segment and Globally (ITT Population)
Description: The mean global BBPS scores and scores by colon segment are presented for the ITT population.
  For each of the 3 colon segments (right, transverse and left colon) the BBPS score ranges from 0 - 3 (worst to best), and was assessed by 3 blinded experts:
  * unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared = 0
  * portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid = 1
  * minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well = 2
  * entire mucosa of colon segment seen well with no residual staining, small fragments of stool and/or opaque liquid = 3.
  The global score is the total of the 3 segment scores ranging from 0 - 9 (worst to best). Reconciled scores were based on 3 blinded reviews. Results of analysis for the PP population for right + transverse colon segments presented separately.
Time Frame: Colonoscopy was performed on Day 2.
Population: The ITT population consisted of all randomised patients who received even a partial dose of study treatment. Patients were assessed according to the randomised treatment, regardless of treatment received. Only patients with data available are included.
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Fortrans®: Patients were randomised to receive an oral split-dose of Fortrans® on Day 1 and Day 2. The first dose was taken the evening of Day 1 before the colonoscopy and the second dose was taken 10 - 12 hours after the evening dose on the day of the colonoscopy. Colonoscopy was performed on Day 2 at least 3 hours and no more than 6 hours after the last dose of Fortrans®.
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 140 | 142
units on a scale
  Right Colon BBPS Score | 2.56 (0.58) | 2.42 (0.62)
  Transverse Colon BBPS Score | 2.78 (0.43) | 2.67 (0.52)
  Left Colon BBPS Score | 2.84 (0.39) | 2.78 (0.48)
  Global BBPS Score | 8.17 (1.21) | 7.86 (1.39)
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; Treatment difference for Right Colon BBPS Score; Test type: Superiority; p = 0.0249, ANOVA; A 2-way analysis of variance model (ANOVA) with covariates for centre, age group (≤65; >65), gender and IBD status was used; Adjusted difference = 0.15, 95% CI 2-sided [0.02 to 0.28]
Statistical Analysis 2: Comparison: Eziclen vs Fortrans®; Treatment difference for Transverse Colon BBPS Score; Test type: Superiority; p = 0.0382, ANOVA; A 2-way ANOVA with covariates for centre, age group (≤65; >65), gender and IBD status was used; Adjusted difference = 0.11, 95% CI 2-sided [0.01 to 0.22]
Statistical Analysis 3: Comparison: Eziclen vs Fortrans®; Treatment difference for Left Colon BBPS Score; Test type: Superiority; p = 0.2538, ANOVA; A 2-way ANOVA with covariates for centre, age group (≤65; >65), gender and IBD status was used; Adjusted difference = 0.06, 95% CI 2-sided [-0.04 to 0.16]
Statistical Analysis 4: Comparison: Eziclen vs Fortrans®; Treatment difference for Global BBPS Score; Test type: Superiority; p = 0.0256, ANOVA; A 2-way ANOVA with covariates for centre, age group (≤65; >65), gender and IBD status was used; Adjusted difference = 0.33, 95% CI 2-sided [0.04 to 0.62]

3. Secondary Outcome: Mean BBPS Score for Right Colon and Transverse Colon Segment (PP Population)
Description: The mean colon segment BBPS scores for the Right Colon and Transverse Colon segments for the PP population are presented.
  For each of the colon segments (right and transverse colon) the BBPS score ranges from 0 - 3 (worst to best), and was assessed by 3 blinded experts as follows:
  * unprepared colon segment with mucosa not seen due to solid stool that cannot be cleared = 0
  * portion of mucosa of the colon segment seen, but other areas of the colon segment not well seen due to staining, residual stool and/or opaque liquid = 1
  * minor amount of residual staining, small fragments of stool and/or opaque liquid, but mucosa of colon segment seen well = 2
  * entire mucosa of colon segment seen well with no residual staining, small fragments of stool and/or opaque liquid = 3.
  Reconciled scores were based on the 3 blinded reviews.
Time Frame: Colonoscopy was performed on Day 2.
Population: The PP population consisted of all randomised patients who received the preparation of study treatment (whether complete or partial), who underwent the colonoscopy procedure and for whom no protocol violation occurred until colonoscopy. Patients were assessed according to the randomised treatment, regardless of treatment received.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 139 | 135
units on a scale
  Right Colon BBPS Score | 2.55 (0.58) | 2.46 (0.56)
  Transverse Colon BBPS Score | 2.78 (0.43) | 2.70 (0.46)
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; Treatment difference for Right Colon BBPS Score (per protocol population); Test type: Superiority; p = 0.0840, ANOVA; A 2-way ANOVA with covariates for centre, age group (≤65; >65), gender and IBD status was used; Adjusted difference = 0.11, 95% CI 2-sided [-0.02 to 0.24]
Statistical Analysis 2: Comparison: Eziclen vs Fortrans®; Treatment difference for Transverse Colon BBPS Score (per protocol population); Test type: Superiority; p = 0.1320, ANOVA; A 2-way ANOVA with covariates for centre, age group (≤65; >65), gender and IBD status was used; Treatment difference = 0.08, 95% CI 2-sided [-0.02 to 0.18]

4. Secondary Outcome: The Percentage of Patients in Whom Lesions Were Detected.
Description: The percentage of patients for whom polyps, adenomas and other lesions were detected during the colonoscopy are presented.
Time Frame: Colonoscopy was performed on Day 2.
Population: The ITT population consisted of all randomised patients who received even a partial dose of study treatment. Patients were assessed according to the randomised treatment, regardless of treatment received. Percentages are calculated based on the overall ITT population.
Measure: Number; unit: percentage of participants
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 146 | 148
percentage of participants
  Polyps detected | 27.4 | 33.8
  Adenomas detected | 20.5 | 18.9
  Other lesions detected | 15.1 | 16.9
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; Treatment difference for detection of polyps; Test type: Superiority; p = 0.2199, Regression, Logistic; A multivariate logistic regression model, adjusted on centre, age class (≤65; >65), gender and IBD status was used; Adjusted difference = -6.94, 95% CI 2-sided [-17.53 to 3.64]
Statistical Analysis 2: Comparison: Eziclen vs Fortrans®; Treatment difference for detection of adenomas; Test type: Superiority; p = 0.6325, Regression, Logistic; A multivariate logistic regression model, adjusted on centre, age class (≤65; >65), gender and IBD status was used; Adjusted difference = 1.87, 95% CI 2-sided [-6.25 to 9.99]
Statistical Analysis 3: Comparison: Eziclen vs Fortrans®; Treatment difference for detection of other lesions; Test type: Superiority; p = 0.7086, Regression, Logistic; A multivariate logistic regression model, adjusted on centre, age class (≤65; >65), gender and IBD status was used; Adjusted difference = -1.55, 95% CI 2-sided [-9.64 to 6.54]

5. Secondary Outcome: The Percentage of Patients for Whom the Colonoscopy Was Completed
Description: The percentage of patients for whom a total colonoscopy could be completed is presented.
Time Frame: Colonoscopy was performed on Day 2.
Population: The ITT population consisted of all randomised patients who received even a partial dose of study treatment. Patients were assessed according to the randomised treatment, regardless of treatment received.
Measure: Number; unit: percentage of participants
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 146 | 148
percentage of participants | 96.6 | 97.3
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; Test type: Superiority; p = 0.9927, Regression, Logistic; A multivariate logistic regression model, adjusted on centre, age class (≤65; >65), gender and IBD status was used; Adjusted difference = 0.01, 95% CI 2-sided [-3.12 to 3.14]

6. Secondary Outcome: Mean Colonoscopy Duration
Description: The mean colonoscopy duration per treatment group is presented. The duration of colonoscopy was defined as the time from colonoscopy insertion to the time to reach the caecum in minutes.
Time Frame: Colonoscopy was performed on Day 2.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 141 | 144
minutes | 9.80 (6.93) | 10.03 (6.87)
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; Test type: Superiority; p = 0.7039, ANOVA; A 2-way ANOVA with covariates for centre, age group (≤65; >65), gender and IBD status was used; Adjusted difference = -0.30, 95% CI 2-sided [-1.88 to 1.27]

7. Secondary Outcome: Investigator Satisfaction as Determined by Mean Likert Scale Score for Global Evaluation
Description: Investigator satisfaction with the procedure was measured by the mean Likert scale score for global evaluation by the investigator.
  The Likert scale consists of 5 points, and ranges from 0 (poor cleansing) to 4 (excellent cleansing) as follows:
  * presence of faeces and soiled fluid: investigation could not be reliably performed = 0
  * presence of faecal material and of unclear fluid, with negative effect on the reliability of the investigation = 1
  * brown liquid, no solid faecal material, presence of unclear residual fluid that could be aspirated: no effect on the reliability of the investigation = 2
  * absence of solid faecal material, presence of clear residual fluid = 3
  * no faecal material, no residual fluid, empty colon = 4.
Time Frame: Colonoscopy was performed on Day 2.
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 145 | 148
units on a scale | 3.03 (0.61) | 2.93 (0.72)
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; Test type: Superiority; p = 0.1891, ANOVA; A 2-way ANOVA with covariates for centre, age group (≤65; >65), gender and IBD status was used; Adjusted difference = 0.10, 95% CI 2-sided [-0.05 to 0.25]

8. Secondary Outcome: Evaluation of Patient Compliance as Determined by the Percentage of Patients Who Consumed All the Planned Volume of Study Treatment
Description: Patient compliance was evaluated based on the percentage of patients who consumed all the planned volume of the study treatment.
  A patient was considered compliant with the instructions of use provided in the prescription if he/she drank the whole preparation and any required further fluid intake. The percentage of compliant patients is presented.
Time Frame: Study treatment was administered as a split-dose on Days 1 and 2.
Population: as for outcome 5
Measure: Number; unit: percentage of participants
Arm/Group | Eziclen | Fortrans®
Number analyzed (Participants) | 146 | 148
percentage of participants | 96.6 | 84.5
Statistical Analysis 1: Comparison: Eziclen vs Fortrans®; Test type: Superiority; p = 0.0011, Regression, Logistic; A multivariate logistic regression model, adjusted on centre, age class (≤65; >65), gender and IBD status was used; Adjusted difference = 13.35, 95% CI 2-sided [6.37 to 20.32]

ADVERSE EVENTS:
Time Frame: Treatment emergent adverse events (TEAEs) were collected from Day 1 up to 30 +/- 3 days after colonoscopy (approximately 1 month).
Description: AEs were actively collected by the investigator and patients were instructed to contact the investigator if they experienced any AEs. The safety population consisted of all randomised patients who received even a partial dose of study treatment. Patients were analysed according to the actual treatment received.
Arm/Group | Eziclen | Fortrans®
All-Cause Mortality (participants affected / at risk) | 0/147 | 0/147
Serious Adverse Events (participants affected / at risk) | 1/147 | 0/147
Other Adverse Events (participants affected / at risk) | 101/147 | 81/147
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eziclen (N=147) | Fortrans® (N=147)
Proctitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Eziclen (N=147) | Fortrans® (N=147)
Nausea (Gastrointestinal disorders) | 41 (66) | 19 (25)
Abdominal distension (Gastrointestinal disorders) | 27 (38) | 19 (26)
Abdominal discomfort (Gastrointestinal disorders) | 13 (21) | 13 (16)
Abdominal pain (Gastrointestinal disorders) | 11 (15) | 9 (9)
Hyperuricaemia (Metabolism and nutrition disorders) | 18 (20) | 24 (25)
Hyperbilirubinaemia (Hepatobiliary disorders) | 10 (11) | 10 (10)

LIMITATIONS AND CAVEATS:
The differences in the Safety and ITT populations were due to 3 drug administration deviations. 2 patients initially randomized in the Fortrans® group received Eziclen and 1 patient initially randomized in the Eziclen group received Fortrans® .

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
No publication of the Study Results shall be made without Sponsor's prior written approval. If a multi-centre publication is not submitted to a journal within 24 months after study conclusion at all sites the PI may individually publish results from the Institution Site subject to Sponsor's prior approval. Sponsor to be provided with final version of any abstract/presentation/paper prior to disclosure to provide scientific comments within 2 weeks for abstract/presentation or 6 weeks for article.